CLINICAL TRIAL: NCT07203274
Title: The Role of Janus Kinase (JAK) and Voltage-gated Sodium Channels (Nav) on Pain and Itch Sensitivity in Healthy Volunteers
Brief Title: The Role of Janus Kinase (JAK) and Voltage-gated Sodium Channels (Nav) on Pain and Itch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20240054
Record Dates: First submitted 2025-05-28; First posted 2025-10-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Itchiness
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Intervention Model Description: In each participant, the four different creams will be applied in a randomized position. After the cream removal, itch will be induced using histamine in one session and cowhage in the other session.
Masking Description: The participant will be blinded about which cream is applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cream application (Experimental): This subproject will be conducted in two sessions one week apart. Each session will last approximately 4-5 hours. In each forearm of the participant, two 4x4 cm areas will be selected as Area of Interest (AOI). In these selected areas, the four different creams will be applied in randomized position for 1 hour. After the cream removal, itch will be induced using histamine in one session and cowhage in the other session (the order of histamine and cowhage will be randomized). During the application of the substances, the itch/pain elicited will be monitored for 10 minutes using a VAS (Visual analog scale). After the removal of the substances, measurements of SBP, MEI, PTT MPT, MPS, and thermal sensitivity will be conducted.
  Interventions: Drug: Delgocitinib cream; Drug: lidocaine cream; Combination Product: Lidocaine+Delgocitinib; Drug: Vehicle (placebo); Other: Histamine Dihydrochloride (HDC); Other: Cowhage (Mucuna Pruriens)

INTERVENTIONS:
Drug: Delgocitinib cream — Delgocitinib cream
Drug: lidocaine cream — Lidocaine cream
Combination Product: Lidocaine+Delgocitinib — The two cream will me mixed togheter
Drug: Vehicle (placebo) — Vehicle Cream
Other: Histamine Dihydrochloride (HDC) — One drop of histamine will be applied on the selected areas and pierced with a lancet
Other: Cowhage (Mucuna Pruriens) — About 30 spicules will be applied on the selected areas and inserted manually

SUMMARY:
It is well known that itch and pain have many communalities in terms of pathways and molecules involved. Therefore, it is very important to investi-gate different substances that work against both pain and itching. The substances delgocitinib and lidocaine have both been shown to relieve various types of pain. We therefore assume that these creams will be also able to relieve itching. The purpose of this trial experiment is therefore to investigate the effect of delgocitinib, lidocaine and their combination on experimentally induced itching.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

  * 18-60 years
  * Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation

  * Drug addiction defined as any use of cannabis, opioids, or other drugs that may cause addiction.
  * Previous or current history of neurological, dermatological (e.g., AD, psoriasis, etc.), immunological, musculoskeletal, cardiac disorder or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
  * Moles, wounds, scars, or tattoos in the area to be treated or tested
  * Current use of medications that may affect the trial such as antihistamines and painkillers
  * use of antihistamines should be discontinued 72 hours before the experiment and all topical agents and emollients should be discontinued 24 hours before the experiment).
  * Use of systemic and topical corticosteroids
  * Previous traumatic experience of an electrical accident
  * Application of moisturizing lotion of the volar site of the forearms (24 hours before study start)
  * Skin diseases
  * Consumption of alcohol or painkillers 24 hours before the study days and between these
  * Acute or chronic pain and itch
  * Known allergy/intolerance to lidocaine/phenytoin/mepyramine
  * Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
  * Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring itch by computerized Visual Analog Scale Scoring | Day 1
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring itch by computerized Visual Analog Scale Scoring | Day 2
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Superficial blood perfusion | Day 1
Superficial blood perfusion | Day 2

SECONDARY OUTCOMES:
Mechanically evoked itch (MEI) | Day 1
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch (MEI) | Day 2
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Perception threshold tracking model (PTT) | Day 1
Perception threshold tracking model (PTT) | Day 2
Mechanical Pain Thresholds (MPT) | Day 1
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Thresholds (MPT) | Day 2
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Day 1
  This test is conducted with the same pinprick set used to test the MPT.
Mechanical Pain Sensitivity (MPS) | Day 2
  This test is conducted with the same pinprick set used to test the MPT.
Warm Detection Thresholds (WDT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 2
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Thresholds (CDT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Thresholds (CDT) | Day 2
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 2
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Day 2
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 2
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain Faculty of Medicine, Aalborg University Selma Lagerløfs Vej 249 9260 Gistrup, Denmark, Gistrup, Denmark